CLINICAL TRIAL: NCT03048175
Title: Systemic Inflammation After Wisdom Tooth Removal: a Case-control Study
Brief Title: Acute Inflammation After Wisdom Tooth Removal
Acronym: OTTO-SYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Associate Professor, University of Pisa
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2198
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Tooth Impacted
Keywords: C-reactive protein; Systemic inflammation; Third molar; Wisdom tooth
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: Case-control intervention trial: cases are treated for pathology. Controls do not have pathology.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Code was assigned to each participant. No info on whether they belong to cases or control was given to researchers and statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases: wisdom tooth pathology (Experimental): Subjects affected by bilateral wisdom tooth pathology, undergoing surgical removal
  Interventions: Procedure: Wisdom tooth removal
- Controls: no wisdom tooth pathology (No Intervention): Subjects showing agenesia/previous extraction/no symptoms of the lower third molars.

INTERVENTIONS:
Procedure: Wisdom tooth removal — After inferior dental and buccal nerve anesthesia a triangular full thickness flap with releasing incision on the mesio-buccal aspect of the second molar is designed. Ostectomy is then performed and tooth is sectioned and gently elevated. Once all the tooth components are extracted, the socket is carefully inspected and flap is sutured with interrupted sutures.
  Arms: Cases: wisdom tooth pathology

SUMMARY:
Third molar (wisdom teeth) extraction is one of the most frequent intervention in dentistry. Nevertheless, little is known about the level of general body inflammation of subjects with impacted or semi-impacted third molars. Moreover, The possible effects of surgical removal of wisdom teeth on the overall health are not known.

Thus, a study in which 40 subjects has been designed. Twenty subjects were affected by bilateral wisdom tooth pathology necessitating for extraction of both teeth. Control group comprised 20 subjects with absence of wisdom teeth or completely erupted wisdom teeth without pathology associated to or history of previous extraction of both wisdom teeth.

In both groups a medical and dental examination will be performed at the baseline and 3 months after baseline for the control group or after the second third molar extraction in the control group. Blood will be also withdrawn to assess systemic inflammation and other systemic parameters.

Parameter were evaluated via high sensitive c reactive protein (CRP), lipids, fibrinogen, oxidative stress and endothelial function analysis.

DETAILED DESCRIPTION:
Third molar extraction is one of the most frequent intervention in dentistry. Nevertheless, little is known about the systemic aspect of subjects with impacted or semi-impacted third molars and the possible effects of surgical removal on their systemic parameters. A case-control study of 40 subjects has been designed to evaluate i) the overall systemic inflammation and metabolism of subjects with bilateral third molars compared to subjects with no third molars and ii) the effect of bilateral removal in the immediate and medium postsurgical period. Systemic parameters are evaluated via high sensitive c reactive protein (CRP), lipids, fibrinogen, oxidative stress and endothelial function analysis.

ELIGIBILITY:
Inclusion Criteria:

* cases: bilateral wisdom tooth pathology.
* control: agenesia/previous extraction/no symptoms of the lower third molars.

Exclusion Criteria:

* younger than 18 years and older than 65 years;
* pregnant or lactating females;
* females using contraceptive methods;
* suffering from any systemic illness;
* undergoing any pharmacological treatment within 30 days prior to the inclusion
* patients affected by periodontal disease (radiographic diagnosis of vertical bone defects or bone resorption equal to 20% of the root length);
* patients with periapical and periradicular radiolucent areas X-ray detectable;
* patients unable to participate to study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04-19 (Actual); Primary Completion 2009-06-15 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in C-reactive protein (CRP) | baseline, 24 and three months after the second extraction
  High-Sensitive plasmatic C-reactive protein

SECONDARY OUTCOMES:
Changes in plasma malondialdehyde (MDA) | baseline, 24 and three months after the second extraction
  plasma malondialdehyde
Changes in lipoperoxides (LOOH) | baseline, 24 and three months after the second extraction
  lipoperoxides levels in plasma
Changes in ferric-reducing antioxidant power (FRAP) | baseline, 24 and three months after the second extraction
  FRAP levels in plasma
Changes in endothelial flow-mediated dilation (FMD) calculated as maximal percentual increase in diameter of the blood vessel above baseline | baseline, 24 and three months after the second extraction
  Endothelium-dependent response of the brachial artery in response to increased blood flow by high resolution ultrasound with a 7.5 MHz linear array transducer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graziani F, D'Aiuto F, Gennai S, Petrini M, Nisi M, Cirigliano N, Landini L, Bruno RM, Taddei S, Ghiadoni L. Systemic Inflammation after Third Molar Removal: A Case-Control Study. J Dent Res. 2017 Dec;96(13):1505-1512. doi: 10.1177/0022034517722775. Epub 2017 Jul 31. PMID 28759304